CLINICAL TRIAL: NCT00965497
Title: An Open-label, 8- Week, Flexible Dose Trial of Escitalopram (Lexapro®) in Comorbid Major Depression With Amyotrophic Lateral Sclerosis and Multiple Sclerosis
Brief Title: Escitalopram (Lexapro) for Depression MS or ALS
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of South Carolina (Other)
Responsible Party: Principal Investigator, Meera Narasimhan, Professor, University of South Carolina
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Pro00003013
Record Dates: First submitted 2009-08-07; First posted 2009-08-25 (Estimated); Results first posted 2011-09-07 (Estimated); Last update posted 2019-05-01 (Actual); Status verified 2011-08

CONDITIONS: Major Depression; Multiple Sclerosis; Amyotrophic Lateral Sclerosis
Keywords: Amyotrophic Lateral Sclerosis; ALS; Multiple Sclerosis; MS; Major Depression; Depression; Major Depressive Disorder; antidepressants; Escitalopram; Lexapro
MeSH Terms: conditions — Depressive Disorder, Major; Multiple Sclerosis; Amyotrophic Lateral Sclerosis; Depression | interventions — Escitalopram

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Escitalopram (Experimental): All patients will receive escitalopram 20 mg daily.
  Interventions: Drug: escitalopram

INTERVENTIONS:
Drug: escitalopram — After confirmation of diagnoses and safety screening escitalopram will be started at 10 mg per day and augmented weekly in 10 mg per day increments, the maximum dose being 20 mg per day. The dose will be titrated upward or downward based on clinical response and tolerability. No other psychotropic medications will be permitted during the study. Medications for coexisting medical problems (e.g. hypertension) will be permitted. Study visits will include weekly visits for first 2 weeks and biweekly visits for next 6 weeks. Medications will be dispensed weekly or biweekly and the participants will be followed for 8 weeks.
  Other Names: Lexapro

SUMMARY:
The purpose of this study is to see if escitalopram (Lexapro) improves symptoms of major depressive disorder in patients who have ALS or MS.

DETAILED DESCRIPTION:
This eight-week study aims to assess the effectiveness and tolerability of escitalopram in improving symptoms of Major Depression in patients with Amyotrophic Lateral Sclerosis (ALS) or Multiple Sclerosis (MS) as measured by the HAM-D. In addition, the study will assess improvement in the quality of life in patients with Major Depression and ALS or MS.

ELIGIBILITY:
Inclusion Criteria:

* Patients between 18 and 70 years of age with documented ALS or MS,
* DSM-IV episode of non-psychotic Major Depression,
* ≥14 score on the 17-item HAM-D,
* Ability to give informed consent.

Exclusion Criteria:

* History of psychotic disorders,
* Psychotic depression,
* Bipolar depression,
* Suicide risk,
* History of substance abuse in the previous 6 months,
* History of unstable medical disorders,
* Pregnancy or planning for pregnancy,
* Severity of ALS or MS that limits participating in the study protocol.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2009-07; Primary Completion 2010-03 (Actual); Study Completion 2010-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Meera Narasimhan, MD, Principal Investigator — University of South Carolina School of Medicine
Locations (1):
- University of South Carolina School of Medicine, Columbia, South Carolina, United States

REFERENCES:
- [Background] Cohen SR, Mount BM, Strobel MG, Bui F. The McGill Quality of Life Questionnaire: a measure of quality of life appropriate for people with advanced disease. A preliminary study of validity and acceptability. Palliat Med. 1995 Jul;9(3):207-19. doi: 10.1177/026921639500900306. PMID 7582177
- [Background] Ganzini L, Johnston WS, Hoffman WF. Correlates of suffering in amyotrophic lateral sclerosis. Neurology. 1999 Apr 22;52(7):1434-40. doi: 10.1212/wnl.52.7.1434. PMID 10227631

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruited through local neurology groups and ALS and MS support groups. No subjects with ALS were recruited.
Pre-assignment Details: Patients switched from another antidepressant to escitalopram were either cross-titrated to escitalopram over 1 week or went through 3 day washout before starting escitalopram. Subjects with uncontrolled medical conditions (i.e., uncontrolled hypertension)were excluded.
Groups:
- Open-label, Single Arm: All patients will receive the intervention
Period: Overall Study
Arm/Group | Open-label, Single Arm
Started | 14
Completed | 13
Not Completed | 1
Not completed — Physician Decision | 1

BASELINE CHARACTERISTICS:
Arm/Group | Open-label, Single Arm
Number analyzed (Participants) | 14
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 14
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12
  Male | 2
Region of Enrollment [Number; unit: participants]
  United States | 14

OUTCOME MEASURES:

1. Primary Outcome: Hamilton Depression Scale (HAM-D 17).
Description: Hamilton Depression Rating Scale-17 (HAM-D) is a 17-item observer rated scale that measures depressive symptoms. Items are rated 0 (no symptoms)-4 ( most severe symptoms. Possible minimum and maximum scores range is 0-50. total score indications: 0-7 = Normal; 8-13 = Mild Depression; 14-18 = Moderate Depression; 19-22 = Severe Depression and ≥ 23 = Very Severe Depression.
Time Frame: 8 weeks
Population: Intention to Treat
Measure: Median (Standard Deviation); unit: depression severity
Groups:
- Escitalopram: One-arm study of escitalopram 20 mg daily
Arm/Group | Escitalopram
Number analyzed (Participants) | 13
depression severity | 15 (7)
Statistical Analysis 1: Comparison: Escitalopram; There were 13 people that completed so there truly was no power to detect true differences; therefore only trends can be discussed; Test type: Superiority or Other; p = 0.01, t-test, 2 sided; Mean Difference (Final Values) = 95

2. Secondary Outcome: McGill Quality of Life Scale (MQOL)
Description: McGill Quality of Life Scale is a a 20-item scale measuring quality of life in chronic and end of life conditions. MQOL is self-reported with a 2-day time frame. Items are scored 0 (worst) to 10 (excellent)on five domains (physical well-being, physical symptoms, psychological, existential, and support). An overall index score can be calculated from the means of the five sub-scales measuring quality of life from 0 (poor) to 10 (excellent).
Time Frame: 8 weeks
Measure: Mean (Full Range); unit: quality of life
Arm/Group | Escitalopram
Number analyzed (Participants) | 13
quality of life | 5 [0 to 10]

ADVERSE EVENTS:
Arm/Group | Open-label, Single Arm
Serious Adverse Events (participants affected / at risk) | 0/14
Other Adverse Events (participants affected / at risk) | 5/14
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Open-label, Single Arm (N=14)
Nausea vomiting and diarrhea (Gastrointestinal disorders) | 5 (5)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No